CLINICAL TRIAL: NCT05383170
Title: A Phase 1b/2a, Open-Label, Multi-Center Study of CyPep-1 in Combination With Pembrolizumab to Evaluate the Efficacy and Safety of CyPep-1 in Patients With Advanced or Metastatic Head and Neck Squamous Cell Carcinoma (HNSCC), Melanoma, or Triple-Negative Breast Cancer (TNBC) (CATALYST)
Brief Title: A Study to Evaluate the Safety and Efficacy of CyPep-1 in Combination With Pembrolizumab for the Treatment of Advanced or Metastatic Cancers
Acronym: Catalyst
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cytovation AS (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CYP003; 2021-006804-34 (EudraCT Number); KEYNOTE-D11 (Other: Merck Sharp & Dohme LLC); MK-3475-D11 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2022-05-03; First posted 2022-05-20 (Actual); Results first posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-10

CONDITIONS: Advanced Head and Neck Squamous Cell Carcinoma; Advanced Breast Cancer; Advanced Melanoma
Keywords: Cancer; Tumour; Oncology; Immunotherapy; Oncolytic; CD8; Intratumoral; Neoplasm; itRECIST
MeSH Terms: conditions — Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: advanced or metastatic HNSCC (Experimental): The safety and tolerability of CyPep-1 in combination with pembrolizumab will be evaluated in a cohort of 30 subjects in total with advanced or metastatic HNSCC. CyPep-1 will be administered every 2 weeks (Q2W) and pembrolizumab will be administered following a Q6W schedule as per standard of care (SoC).
  Interventions: Drug: CyPep-1; Drug: Pembrolizumab 25 MG/ML [KEYTRUDA®]
- Arm B: advanced or metastatic melanoma (Experimental): The safety and tolerability of CyPep-1 in combination with pembrolizumab will be evaluated in a cohort of 30 subjects in total with advanced or metastatic melanoma. CyPep-1 will be administered every 2 weeks (Q2W) and pembrolizumab will be administered following a Q6W schedule as per standard of care (SoC).
  Interventions: Drug: CyPep-1; Drug: Pembrolizumab 25 MG/ML [KEYTRUDA®]
- Arm C: advanced or metastatic TNBC (Experimental): The safety and tolerability of CyPep-1 in combination with pembrolizumab will be evaluated in a cohort of 30 subjects in total with advanced or metastatic TNBC. CyPep-1 will be administered every 2 weeks (Q2W) and pembrolizumab will be administered following a Q6W schedule as per standard of care (SoC).
  Interventions: Drug: CyPep-1; Drug: Pembrolizumab 25 MG/ML [KEYTRUDA®]

INTERVENTIONS:
Drug: CyPep-1 — Intratumoral injection
Drug: Pembrolizumab 25 MG/ML [KEYTRUDA®] — IV infusion
  Other Names: KEYTRUDA®

SUMMARY:
This Phase 1b/2a study will assess the efficacy, safety, and pharmacodynamics of CyPep-1 when administered directly into measurable tumor lesions in combination with the anti-PD-1 antibody pembrolizumab. Additionally, the study will assess anti-tumor effects of CyPep-1 on injected lesions and non-injected target lesions identified at baseline, as well as local and systemic immunological effects of CyPep-1 in combination with pembrolizumab.

DETAILED DESCRIPTION:
Treatment with immune modulating agents may result in long lasting anti-tumor responses in patients with cancer. However, only a subset of patients obtains durable remission. Treatment strategies that aim at recruiting tumor antagonizing cellular components of the immune system holds great promise.

CyPep-1 is a chemically synthesized peptide with oncolytic properties. It selectively targets cancer cells based on their altered molecular composition, and removes the surrounding cell membrane. This releases tumor neoantigens to the microenvironment and potentially induces an anti-tumour immune response.

Preclinical studies show that CyPep-1 can synergize with anti-PD-1 antibody treatment in terms of decreased tumor volumes and prolonged Overall Survival (OS), highlighting the possible clinical utility of CyPep-1 in the combination setting with ICIs.

This is an open-label, multi-center, non-randomized Phase 1b/2a study. The Phase 1b portion of the study (ie, the first 6 patients enrolled) will confirm the recommended CyPep-1 dose of 20 mg every 2 weeks (Q2W) in combination with pembrolizumab 400 mg every 6 weeks (Q6W). The patients from the Phase 1b portion will continue to the Phase 2a portion of the study (approximately 90 patients in total will be enrolled, with 30 patients per arm). The Phase 2a portion of the study will have 3 arms including patients with advanced or metastatic HNSCC, melanoma, or TNBC and will assess the efficacy, safety, and pharmacodynamics of CyPep-1 (20 mg Q2W) when administered directly into measurable tumor lesions in combination with the anti-programmed cell death protein 1 (PD-1) antibody pembrolizumab (400 mg Q6W).

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria

1. Is 18 years of age or older on the day of signing informed consent;
2. Provides written informed consent and is able to comply with study procedures and assessments;
3. Has measurable disease as determined by the Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1;
4. Has at least 1 non-ulcerated, measurable, and accessible lesion for intra-tumoral (IT) injection with a maximum diameter of 5 cm;
5. Is able to provide tissue from a core or excisional biopsy at screening or has an acceptable stored tumor sample available that was collected within 90 days prior to screening;
6. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
7. Has a life expectancy >=3 months, as determined by the Investigator;
8. Female patients of non-childbearing potential must be either surgically sterile (hysterectomy, bilateral tubal ligation, salpingectomy, and/or bilateral oophorectomy at least 26 weeks before screening), post-menopausal, defined as spontaneous amenorrhea for at least 2 years, or with follicle-stimulating hormone in the post-menopausal range at screening;
9. Female patients of childbearing potential (defined as <2 years after last menstruation or not surgically sterile) must have a negative serum pregnancy test at screening and agree to use a highly effective method for contraception from the time of signing the ICF until at least 120 days after the last administration of CyPep-1.
10. If a male patient is able to father children, he must agree to use 2 acceptable methods of contraception throughout the study (eg, condom plus permicidal gel). Sperm donation is not recommended from the time of signing the ICF until at least 120 days after the last administration of CyPep-1
11. Has adequate organ function. Specimens must be collected within 72 hours prior to the start of study treatment at Cycle 1 Visit 1.

Inclusion Criteria for Arm A

Patients who meet all of the general Inclusion Criteria and the following additional criteria will be eligible for inclusion in Arm A:

1. Have histologically confirmed diagnosis of HNSCC (including nasopharyngeal squamous cell carcinoma);
2. Have advanced or metastatic HNSCC incurable by standard of care therapies; and
3. Have failed or progressed on or after prior platinum-based therapy OR has failed or progressed on or after treatment with a checkpoint inhibitor administered either as monotherapy or in combination with other therapies (if immune checkpoint inhibitor [ICI] eligible based on programmed cell death ligand 1 [PD-L1] status).

Inclusion Criteria for Arm B

Patients who meet all of the general Inclusion Criteria and the following additional criteria will be eligible for inclusion in Arm B:

1. Have histologically confirmed diagnosis of malignant melanoma;
2. Do not have uveal melanoma
3. Have advanced or metastatic melanoma incurable by standard of care therapies;
4. Have received a combination of a BRAF inhibitor and a MEK inhibitor if diagnosed with a BRAF mutated melanoma and if clinically indicated; and
5. Have failed or progressed on or after treatment with a checkpoint inhibitor administered either as monotherapy or in combination with other checkpoint inhibitors or other therapies.

Inclusion Criteria for Arm C

Patients who meet all of the general Inclusion Criteria and the following additional criteria will be eligible for inclusion in Arm C:

1. Have histologically confirmed diagnosis of TNBC;
2. Have advanced or metastatic TNBC incurable by standard of care therapies;
3. Have received sacituzumab govitecan chemotherapeutic treatment if clinically indicated; and
4. Have failed or progressed on or after treatment with a checkpoint inhibitor administered either as monotherapy or in combination with other therapies (if ICI eligible based on PD-L1 status) OR have received prior systemic therapy with either an anthracycline- or taxane-containing regimen (if ICI non-eligible based on PD-L1 status).

Exclusion Criteria:

1. Has only non-palpable cutaneous infiltrations (eg, breast cancer cutaneous carcinomatosis);
2. Had anti-cancer therapy within 4 weeks prior to the first dose of CyPep-1 (2 weeks for palliative radiotherapy);
3. Has participated in a clinical trial and received an investigational therapy within 30 days prior to the first dose of CyPep-1;
4. Has received or will receive a live or live attenuated vaccine within 30 days prior to the first dose of CyPep-1; Note: Seasonal flu vaccines that do not contain live vaccine are permitted. Coronavirus Disease 2019 (COVID-19) vaccines are only permitted with documentation of the date of the vaccine if the last dose of vaccine was administered >14 days prior to the first dose of CyPep-1. The COVID-19 booster vaccine must be administered at least 14 days prior to the first dose of CyPep-1 and is not allowed during the first 3 months of the Treatment Period.
5. Has tested positive for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection within 14 days prior to the Screening Visit; Note: Patients who have had a known SARS-CoV-2 infection >14 days prior to the Screening Visit are permitted at Investigator discretion and must present with no symptoms.
6. Has had a major surgical procedure within 14 days prior to the first dose of CyPep-1;
7. Is expected to require a systemic or localized antineoplastic therapy during participation in this study, excluding localized palliative radiotherapy to tumors not selected for evaluation of treatment response; Note: Use of denosumab for patients with bone metastasis is allowed.
8. Is pregnant or breastfeeding;
9. Has clinical evidence of a secondary malignancy actively progressing or requiring active treatment other than curative therapies for early stage (carcinoma in situ or Stage 1) carcinomas or non-melanoma skin cancer;
10. Has had any autoimmune disease requiring immunosuppressive therapy (ie, use of disease modifying agents, corticosteroids, or immunosuppressive drugs) within 2 years prior to the first dose of CyPep-1; Note: Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
11. Has a condition requiring continuous systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive agents within 2 weeks prior to the first dose of CyPep-1. Inhaled, intranasal, or topical (only on areas outside the injected lesion[s]) and physiological replacement doses of up to 10 mg daily prednisone equivalent are permitted in the absence of active autoimmune disease;
12. Has abnormal or clinically significant coagulation parameters as determined by the Investigator (eg, prothrombin time, international normalized ratio, activated partial thromboplastin time) unless patients are on anticoagulants in which case it must be within appropriate clinical levels; Note: Patients who are on anticoagulants must be able to switch to a low molecular weight heparin or equivalent prior to Cycle 1 Day 1 and continue during the Treatment Period.
13. Has a significant history or clinical manifestation of any allergic disorders and/or Quincke's edema (as determined by the Investigator) capable of significantly altering the absorption of drugs, of constituting a risk when taking CyPep-1 or pembrolizumab, or of interfering with the interpretation of the data;
14. Has a known hypersensitivity to any component of CyPep-1 or pembrolizumab;
15. Has a history of adverse reactions from treatment with ICIs, including pembrolizumab, which resulted in discontinuation of ICI or pembrolizumab or has ongoing pembrolizumab-related toxicity event(s) as per treatment-limiting toxicity definitions, except patients with ongoing endocrine disorders that are managed with replacement therapy (ie, hypothyroidism related to prior pembrolizumab treatment);
16. Has an active infection requiring systemic therapy;
17. Has a known history of Hepatitis B or known active Hepatitis C virus infection;
18. Has had radiotherapy within 2 weeks prior to the first dose of CyPep-1, is in recovery from radiation toxicity, or has had radiation pneumonitis;
19. Has a history of non-infectious pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease;
20. Has had a prior allogeneic tissue/solid organ transplant, stem cell, or bone marrow transplant;
21. Has active human immunodeficiency virus (HIV). Patient is eligible when on stable antiretroviral therapy (no change in medication or dose) for at least 4 weeks prior to screening, has confirmed virologic suppression with HIV RNA less than 50 copies/mL or the lower limit of quantification (below the limit of detection) using the locally available assay at the time of screening and for at least 12 weeks prior to screening, and has a cluster of differentiation 4+ T cell count >350 cells/mm3 at screening. HIV-infected patients with a history of Kaposi sarcoma and/or Multicentric Castleman Disease will be excluded;
22. Have 4 or more sites involved, including the primary cancer; Note: A site is defined as an organ (eg, lung, liver, or brain) or a system (eg, lymphatic or central nervous system [CNS]).
23. Has a central nervous system (CNS) metastasis that is symptomatic, progressing, or that requires current therapy (eg, evidence of new or enlarging CNS metastasis, carcinomatous meningitis, or new neurological symptoms attributable to CNS metastasis);
24. Has a QTcF >480 ms at screening, history of long or short QT syndrome, Brugada syndrome, QTc prolongation, or Torsade de Pointes, with the exception of patients with controlled atrial fibrillation, pacemaker, or bundle branch block as the QTc will be prolonged due to the widened QRS;
25. Are an adult under legal protection, are vulnerable, or lack the capacity to give informed consent, such as: persons deprived of liberty by a judicial or administrative decision; adult persons subject to a legal protection measure (under supervision/under guardianship); or persons under a judicial protection measure; or
26. Has a history of or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or make participation in the study not in the best interest of the patient, in the opinion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2024-09-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (6):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City Of Hope, Duarte, California
  - Henry Ford Health System, Detroit, Michigan
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Houston Methodist, Houston, Texas
- France (8):
  - CHRU de Besançon, Besançon
  - Institut Bergonie, Bordeaux
  - CHU Lille, Lille
  - Centre Leon Berard, Lyon
  - AP-HM - Hôpital de la Timone, Marseille
  - Institut Paoli Calmettes, Marseille
  - Hôpital Saint Louis - AP-HP, Paris
  - Institute Gustave Roussy, Villejuif
- Italy (2):
  - Istituto Europeo di Oncologia, Milan
  - Azienda Ospedaliero Universitaria Senese, Siena
- Netherlands (3):
  - NKI/AvL, Amsterdam
  - Maastricht UMC, Maastricht
  - EMC, Rotterdam
- Spain (6):
  - Vall d'Hebron (VHIO), Barcelona
  - Clinica Universidad de Navarra Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Clinica Universidad de Navarra Pamplona, Pamplona
  - Hospital Universitario Virgen Macarena, Seville

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gibney GT, Weiner LM, Atkins MB. Predictive biomarkers for checkpoint inhibitor-based immunotherapy. Lancet Oncol. 2016 Dec;17(12):e542-e551. doi: 10.1016/S1470-2045(16)30406-5. PMID 27924752
- [Background] Herbst RS, Soria JC, Kowanetz M, Fine GD, Hamid O, Gordon MS, Sosman JA, McDermott DF, Powderly JD, Gettinger SN, Kohrt HE, Horn L, Lawrence DP, Rost S, Leabman M, Xiao Y, Mokatrin A, Koeppen H, Hegde PS, Mellman I, Chen DS, Hodi FS. Predictive correlates of response to the anti-PD-L1 antibody MPDL3280A in cancer patients. Nature. 2014 Nov 27;515(7528):563-7. doi: 10.1038/nature14011. PMID 25428504
- [Background] Samstein RM, Lee CH, Shoushtari AN, Hellmann MD, Shen R, Janjigian YY, Barron DA, Zehir A, Jordan EJ, Omuro A, Kaley TJ, Kendall SM, Motzer RJ, Hakimi AA, Voss MH, Russo P, Rosenberg J, Iyer G, Bochner BH, Bajorin DF, Al-Ahmadie HA, Chaft JE, Rudin CM, Riely GJ, Baxi S, Ho AL, Wong RJ, Pfister DG, Wolchok JD, Barker CA, Gutin PH, Brennan CW, Tabar V, Mellinghoff IK, DeAngelis LM, Ariyan CE, Lee N, Tap WD, Gounder MM, D'Angelo SP, Saltz L, Stadler ZK, Scher HI, Baselga J, Razavi P, Klebanoff CA, Yaeger R, Segal NH, Ku GY, DeMatteo RP, Ladanyi M, Rizvi NA, Berger MF, Riaz N, Solit DB, Chan TA, Morris LGT. Tumor mutational load predicts survival after immunotherapy across multiple cancer types. Nat Genet. 2019 Feb;51(2):202-206. doi: 10.1038/s41588-018-0312-8. Epub 2019 Jan 14. PMID 30643254
- [Background] Schumacher TN, Schreiber RD. Neoantigens in cancer immunotherapy. Science. 2015 Apr 3;348(6230):69-74. doi: 10.1126/science.aaa4971. PMID 25838375
- [Background] Snyder A, Makarov V, Merghoub T, Yuan J, Zaretsky JM, Desrichard A, Walsh LA, Postow MA, Wong P, Ho TS, Hollmann TJ, Bruggeman C, Kannan K, Li Y, Elipenahli C, Liu C, Harbison CT, Wang L, Ribas A, Wolchok JD, Chan TA. Genetic basis for clinical response to CTLA-4 blockade in melanoma. N Engl J Med. 2014 Dec 4;371(23):2189-2199. doi: 10.1056/NEJMoa1406498. Epub 2014 Nov 19. PMID 25409260
- [Background] Vesely MD, Schreiber RD. Cancer immunoediting: antigens, mechanisms, and implications to cancer immunotherapy. Ann N Y Acad Sci. 2013 May;1284(1):1-5. doi: 10.1111/nyas.12105. PMID 23651186
- [Background] Zappasodi R, Merghoub T, Wolchok JD. Emerging Concepts for Immune Checkpoint Blockade-Based Combination Therapies. Cancer Cell. 2018 Apr 9;33(4):581-598. doi: 10.1016/j.ccell.2018.03.005. PMID 29634946
- [Background] Seymour L, Bogaerts J, Perrone A, Ford R, Schwartz LH, Mandrekar S, Lin NU, Litiere S, Dancey J, Chen A, Hodi FS, Therasse P, Hoekstra OS, Shankar LK, Wolchok JD, Ballinger M, Caramella C, de Vries EGE; RECIST working group. iRECIST: guidelines for response criteria for use in trials testing immunotherapeutics. Lancet Oncol. 2017 Mar;18(3):e143-e152. doi: 10.1016/S1470-2045(17)30074-8. Epub 2017 Mar 2. PMID 28271869
- [Background] Goldmacher GV, Khilnani AD, Andtbacka RHI, Luke JJ, Hodi FS, Marabelle A, Harrington K, Perrone A, Tse A, Madoff DC, Schwartz LH. Response Criteria for Intratumoral Immunotherapy in Solid Tumors: itRECIST. J Clin Oncol. 2020 Aug 10;38(23):2667-2676. doi: 10.1200/JCO.19.02985. Epub 2020 Jun 18. No abstract available. PMID 32552274

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Phase 2a part of the study was not initiated and the trial was stopped with 6 patients enrolled in Phase 1b and when the Phase 1b portion of the trial had been successfully completed. The decision not to proceed with the Phase 2a part of the trial was taken following a reassessment of target indications for CyPep-1.
Period: Overall Study
Arm/Group | Arm A: Advanced or Metastatic HNSCC | Arm B: Advanced or Metastatic Melanoma | Arm C: Advanced or Metastatic TNBC
Started | 1 | 5 | 0
Completed | 1 | 5 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Phase 1b population of the study which consist of the first 6 patients enrolled. According to the SAP, in general, all summaries will be displayed in Total for Phase 1b. By-arm summaries will not be displayed given the small sample size in Phase 1b.
Groups:
- Phase 1b: Phase 1b population of the study which consist of the first 6 patients enrolled. According to the SAP, in general, all summaries will be displayed in Total for Phase 1b. By-arm summaries will not be displayed given the small sample size in Phase 1b.
Arm/Group | Phase 1b
Number analyzed (Participants) | 6
Age, Customized [Mean (Standard Deviation); unit: years] | 55.7 (10.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
ECOG [Number; unit: participants] — Participants were eligible for the study with an Eastern Cooperative Oncology Group (ECOG) performance status of 0 (fully active, able to carry on all pre-disease performance without restriction) or 1 (restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, eg, light housework, office work).
  participants
    0 | 5
    1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Frequency, and Seriousness of TEAEs
Description: Number of CyPep-1 related TEAEs per grading.
Time Frame: For each subject, from the time of signing the ICF until 30 days (90 days for SAEs) after the last dose of study treatment up to a maximum of 18 months.
Population: as for baseline characteristics
Measure: Number; unit: number of events
Groups:
- Phase 1b: Phase 1 b population
Arm/Group | Phase 1b
Number analyzed (Participants) | 6
number of events
  Grade 1 TEAE | 11
  Grade 2 TEAE | 19
  Grade 3 TEAE | 2
  Grade 4 TEAE | 0
  Grade 5 TEAE | 0

2. Primary Outcome: Incidence of DLTs
Description: Number of DLTs
Time Frame: Initial 6 weeks of treatment.
Population: as for baseline characteristics
Measure: Number; unit: number of DLTs
Arm/Group | Phase 1b
Number analyzed (Participants) | 6
number of DLTs | 1

3. Secondary Outcome: PFS Per RECIST v1.1
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as Increase in the sum of diameters of target lesion(s) identified at baseline to >20% and >5 mm from nadir; unequivocal progression of non-target lesion(s) identified at baseline; and development of new lesion(s).
Time Frame: Up to approximately 18 months
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Phase 1b: Phase 1b population
Arm/Group | Phase 1b
Number analyzed (Participants) | 6
Months | 3.3 [1.9 to 12.0]

4. Secondary Outcome: OS Per RECIST v1.1
Time Frame: Up to approximately 18 months
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1b
Number analyzed (Participants) | 6
Months | 13.4 [4.8 to 14.9]

ADVERSE EVENTS:
Time Frame: For each subject, AEs were collected from the time of signing the ICF until 30 days after the last dose of study treatment and for SAEs from the time of signing the ICF until 90 days after the last dose of study treatment up to a maximum of 18 months.
Arm/Group | Phase 1b
All-Cause Mortality (participants affected / at risk) | 3/6
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b (N=6)
Erysipelas (Infections and infestations) | 1 (1) — LOWER LEFT LIMB ERYSIPELAS
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b (N=6)
Injection site pain (General disorders) | 1 (16)
Asthenia (General disorders) | 2 (2)
Axillary pain (General disorders) | 1 (3)
Chills (General disorders) | 1 (1)
Inkection site paraesthesia (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Phase 1b of the study (ie, the first 6 patients enrolled) was successfully completed per protocol. Following a re-assessment of target indications for CyPep-1, it was decided not to initiate the Phase 2a part of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-11-23): https://cdn.clinicaltrials.gov/large-docs/70/NCT05383170/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-09): https://cdn.clinicaltrials.gov/large-docs/70/NCT05383170/SAP_001.pdf